CLINICAL TRIAL: NCT04199936
Title: Postoperative Electrical Muscle Stimulation (POEMS) to Attenuate Muscle Atrophy
Brief Title: Postoperative Electrical Muscle Stimulation (POEMS)
Acronym: POEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19089; 274048 (Other: IRAS (NHS ethics) application number)
Record Dates: First submitted 2019-11-26; First posted 2019-12-16 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Muscle Atrophy; Postoperative Complications
Keywords: muscle; atrophy; postoperative; disuse; electrical muscle stimulation
MeSH Terms: conditions — Muscular Atrophy; Postoperative Complications; Atrophy

STUDY DESIGN:
Intervention Model Description: Single centre pilot study (randomised internal control trial)
Who Masked: Outcomes Assessor
Masking Description: ultrasound images, DXA scans and EMG results will be given coded labeling by a separate researcher so that investigator analysing results will be blinded to whether scans / EMG results are from intervention or control leg, or start of finish.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMG leg (Experimental): Quadriceps muscle group of postoperative patients randomly selected leg which will undergo electrical muscle stimulation for upto 2 hours on each postoperative day
  Interventions: Device: Electrical Muscle stimulation
- Control leg (No Intervention): Quadriceps muscle group of postoperative patients leg not selected to undergo electrical muscle stimulation

INTERVENTIONS:
Device: Electrical Muscle stimulation — Electrical muscle stimulation
  Arms: EMG leg

SUMMARY:
Patients lose a significant amount of muscle following major abdominal surgery. This is partly due to a catabolic response to the surgical insult and inflammation, but is also probably due to a lack of muscle use secondary to immobility.

This study will aim to assess whether some or even all of postoperative muscle loss in the upper leg muscle group is preventable through electrical muscle stimulation to mimic physical activity.

DETAILED DESCRIPTION:
Following major gastrointestinal surgery patients may loose around 6 % of their skeletal muscle mass in the first 5 days. Whilst some of this loss is as a result of inflammation and starvation, some is due to muscle disuse.

Studies have shown that patients spend 96% of their time being sedentary in the first 5 days following major abdominal surgery and by day 5 are still taking a median of less than 500 steps per day. Studies of healthy volunteers who undergo similar muscle disuse loose approximately 3.5% of skeletal muscle mass over the same time period, indicating that around half of postoperative muscle loss may be due to immobility.

Through the use of electrical muscle stimulation, this study will aim to mimic high levels of exercise in the quadriceps of patients who have undergo major gastrointestinal surgery to see whether this reduces or prevents muscle loss. Patients muscles will be measured using ultrasound and DXA and neuromuscular function will be measured using electromyography.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing major segmental colonic resections or gastric/oesophageal resection
* Sufficient mobility and fitness to complete normal enhanced recovery protocols following surgery
* Ability to give informed consent

Exclusion Criteria:

* Pre-existing neuromuscular disease (including parkinson's disease)
* Pacemaker, implantable cardiac defibrillator or other implanted nerve stimulator device
* Metalwork in both upper legs
* Dementia
* Inability to give informed consent
* Disability preventing normal mobilisation after surgery
* Symptomatic peripheral vascular disease
* Chronic kidney failure of chronic heart failure
* Intubation for > 24 hours post operation
* Return to theatre for surgical complication within first 5 days post operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Vastus Lateralis muscle thickness (cm) | 5 days
  Ultrasound scan (USS) measurement of Vastus Lateralis muscle thickness in stimulated vs non stimulated legs of postoperative patients
Vastus Lateralis muscle fibre length | 5 days
  USS measurement of Vastus Lateralis muscle fibre length in stimulated vs non stimulated legs of postoperative patients
Vastus Lateralis muscle fibre pennation angle | 5 days
  USS measurement of Vastus Lateralis muscle fibre pennation angle in stimulated vs non stimulated legs of postoperative patients
Compound muscle action potentials (CMAP) as measured by surface electromyography | 5 days
  Changes in compound muscle action potentials (as detected by EMG) in stimulated vs non stimulated legs of postoperative patients
Near Fibre Motor Unit Potentials as measured by surface EMG | 5 days
  Changes in motor unit potentials (as detected by EMG) in stimulated vs non stimulated legs of postoperative patients
Motor unit number estimates ((MUNE) as derived from surface EMG analysis) | 5 days
  Changes in MUNE (as derived from surface EMG) in stimulated vs non stimulated legs of postoperative patients

SECONDARY OUTCOMES:
Lean muscle mass | 5 days
  DXA measurements of lean muscle mass in upper leg of stimulated vs non stimulated legs of postoperative patients
Physical activity levels in postoperative patients | 5 days
  Physical activity levels of patients following major gastrointestinal resection surgery on each postoperative day as measured by physical activity monitor
Dietary intake in postoperative patients | 5 days
  Dietary intake of patients following major gastrointestinal resection surgery, as recorded by patient food diary on each postoperative day
Inflammatory response following major abdominal surgery | 5 days
  Inflammatory response (as measured by IL6, TNFalfa and CRP) following major gastrointestinal resection surgery and its correlation with degree of skeletal muscle loss
Acceptability of electrical muscle stimulation in postoperative patients | 5 days
  Patient experience of electrical muscle stimulation following major gastrointestinal resection surgery as measured by visual analogue score measures of patient comfort, distress, harmful effects and enjoyment.

CONTACTS AND LOCATIONS:
Overall Officials: Jon N Lund, MBBCh, DM, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data